CLINICAL TRIAL: NCT01990209
Title: A Phase II Study With Orteronel as Monotherapy in Patients With Metastatic Breast Cancer (MBC) That Expresses the Androgen Receptor (AR)
Brief Title: Orteronel as Monotherapy in Patients With Metastatic Breast Cancer (MBC) That Expresses the Androgen Receptor (AR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 203
Record Dates: First submitted 2013-11-08; First posted 2013-11-21 (Estimated); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Breast Cancer
Keywords: triple-negative breast cancer; orteronel; TAK-700; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — orteronel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orteronel (Experimental): The planned dose of orteronel is 300mg orally (PO) twice daily (BID), for a total daily dose of 600mg.
  Interventions: Drug: Orteronel

INTERVENTIONS:
Drug: Orteronel
  Other Names: Tak-700

SUMMARY:
The androgen receptor (AR) is expressed in 70-90 percent of primary breast tumors and in 75 percent of breast metastases. There is evidence to suggest that Androgen Receptor (AR) may be a target in patients with advanced breast cancer. Breast cancer patients whose tumors do not express the ER, PR or HER2 (triple negative) have very few options for treatment. Orteronel is being developed as an endocrine therapy for relevant hormone-sensitive cancers such as prostrate cancer and breast cancer. Triple-negative metastatic breast cancer patients with AR expression could potentially benefit from anti-androgen therapy like orteronel.

DETAILED DESCRIPTION:
This open-label multicenter study will be conducted in 2 stages.

* Lead-in Phase: The first 6 patients treated will be evaluated to confirm the safety and feasibility of this regimen. After all 6 patients complete at least 4 weeks of treatment, and if no prohibitive toxicities are identified, continuous study treatment will begin.
* Continuous Study Treatment: Patients will continue to be enrolled into both cohorts based on their tumor specificities with an anticipated total of 31 patients in Cohort 1 (ER-/PR-/HER2-/AR+) and an anticipated total of 55 patients in Cohort 2 (ER+ and/or PR+/AR+).

Patients will be evaluated every eight weeks for response to treatment. All patients who respond to treatment (complete response [CR] or partial response [PR]) or have stable disease (SD) will continue to receive orteronel until they develop progressive disease (PD) or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care
2. Patients must have MBC that is measurable or evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Patients with metastases limited to the bones are eligible.
3. Patients with breast tumors that are AR+ (≥10% staining by immunohisto-chemistry). Archived tumor tissue from a primary biopsy or metastatic lesion for centralized determination of AR expression is mandatory. If tissue is limited, the additional correlative testing is optional. If tissue is not available, a patient will not be eligible for enrollment into the study. Patients may enroll based on local laboratory AR assessment, but will need to submit tissue for confirmation at the central laboratory.
4. In addition to having AR+ tumors, patients must fit into 1 of the 2 following categories:

   * Triple negative (ER-/PR-/HER2-) (Note: This group of patients must have received at least 1 and up to 3 prior chemotherapy regimens in the advanced setting.)
   * ER+ and/or PR+ (Note: This group of patients must have received at least 1 and up to 3 prior hormonal therapies and at least one prior chemotherapy treatment in the advanced setting. HER2+ patients in this group must have received a minimum of 2 lines of HER2-directed therapy in the advanced setting.) This group of patients may be pre-menopausal with ovarian suppression or post-menopausal. LHRH agonists maybe used to render ovarian suppression with post-menopausal ranges of estradiol or FSH per institutional guidelines.
5. Female or male patients ≥18 years-of-age
6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
7. Patient has recovered (to Grade ≤1) from all clinically significant toxicities related to prior antineoplastic therapies (with the exception of alopecia)
8. Adequate hematological function, defined as:

   * Absolute neutrophil count (ANC) ≥1.25 x 109/L
   * Platelets ≥75 x 109/L
   * Hemoglobin ≥9 g/dL
9. Adequate liver function, defined as:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the upper limit of normal (ULN), if no liver involvement or ≤5 x ULN with liver involvement
   * Total bilirubin ≤1.5 times the upper limit of normal (ULN) (in patients with known Gilbert Syndrome, a total bilirubin ≤3.0 x ULN, with direct bilirubin ≤1.5 x ULN)
10. Adequate renal function, defined as:

    * Creatinine ≤1.5 x ULN or creatinine clearance ≥40 mL/min as calculated by the Cockcroft-Gault method
11. Screening calculated LVEF of ≥50% by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan
12. Ability to swallow and retain oral medication
13. Male patients (even those post vasectomy) who are willing to use adequate contraceptive measures or abstain from heterosexual intercourse during the entire study treatment period and for 4 months after the last dose of study drug
14. Female patients who are not of child-bearing potential and female patients of child-bearing potential who agree to use adequate contraceptive measures or abstain from heterosexual intercourse during the entire study treatment period and for 4 months after the last dose of study drug, who are not breastfeeding, and who have had a negative serum/urine pregnancy test ≤7 days prior to dosing
15. Life expectancy of ≥3 months
16. Willingness and ability to understand the nature of this study and to comply with the study and follow-up procedures.

Exclusion Criteria:

1. Known hypersensitivity to orteronel or to orteronel excipients, which are listed by formulation in the Investigator Brochure
2. Patients receiving other treatment for breast cancer (includes standard hormonal therapy, chemotherapy, biologic therapy, immunotherapy, or radiation therapy). Patients receiving chronic bisphosphonate or denosumab therapy are eligible.
3. Female patients who are both lactating and breastfeeding or have a positive serum pregnancy test during the screening period.
4. Prior anti-androgen therapy
5. Use of an investigational drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of orteronel, or concurrent treatment. For investigational drugs for which 5 half-lives is less than 21 days, a minimum of 10 days between termination of the investigational drug and administration of orteronel is required.
6. Active brain metastases or leptomeningeal disease. Previously treated brain metastases are allowed provided lesions are stable for at least 3 months as documented by head CT scan or magnetic resonance imaging (MRI) of the brain. Patients must be off steroids, but anti-convulsants are allowed.
7. Patients with known adrenal insufficiency, or patients receiving treatment with ketoconazole, abiraterone, or aminoglutethimide.
8. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
9. Major surgical procedures ≤28 days of beginning study treatment or minor surgical procedures ≤7 days. No waiting is required following port-a-cath placement.
10. Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhea ≥ Grade 2, and malabsorption syndrome).
11. History of myocardial infarction, unstable symptomatic ischemic heart disease, ongoing arrhythmias > Grade 2 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], Version 4.0), thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (eg, pericardial effusion restrictive cardiomyopathy) within 6 months prior to first dose of study drug. Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
12. New York Heart Association (NYHA) Class III or IV heart failure
13. Electrocardiogram (ECG) abnormalities of Q-wave infarction, unless identified 6 or more months prior to screening or QTc Fridericia (F) interval >460 msec
14. Inadequately controlled hypertension (ie, systolic blood pressure [SBP] >160 mmHg or diastolic BP [DBP] >90 mmHg) at 2 separate measurements no more than 60 minutes apart during the Screening visit. Note: patients may be rescreened after adjustment of antihypertensive medications.
15. Known diagnosis of human immunodeficiency virus, active chronic hepatitis B, or C, life-threatening illness unrelated to cancer, or any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with participation in this study
16. Uncontrolled diabetes mellitus. Patients with Type II diabetes are eligible if they require only oral hypoglycemic agents and fasting blood glucose level is ≤120. Patients with Type I diabetes are eligible if their glycosylated hemoglobin (HbAlc) is ≤7.
17. Diagnosis or treatment for another malignancy within 2 years of enrollment, with the exception of adequately treated in-situ carcinoma of the cervix, uteri, basal or squamous cell carcinoma or non-melanomatous skin cancer
18. Inability or unwillingness (including psychological, familial, sociological, or geographical conditions) to comply with study and/or follow-up procedures as outlined in the protocol.
19. Use of a prohibited concomitant medication that cannot be safely discontinued or substituted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-03; Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Burris, III, MD, Study Chair — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Yale School of Medicine, New Haven, Connecticut
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Hope Cancer Center, Terre Haute, Indiana
  - Baptist Hospital East, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Cancer Research Consortium of West Michigan, Grand Rapids, Michigan
  - Cancer Centers of SW Oklahoma, Lawton, Oklahoma
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 71 participants were enrolled
Pre-assignment Details: In this study, the first 6 participants enrolled in cohorts 1 and 2 were evaluated as part of a safety lead-in phase following pre-screening for AR expression. The lead-in did not affect the cohort assignments; the assignment was decided by Inclusion Criteria. After these 6 patients completed at least 4 weeks of treatment without any prohibitive toxicities, the study continued to enroll the rest of the study participants.
Groups:
- Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors: Patients with estrogen receptor-negative (ER-)/progesterone receptor negative (PR-)/ human epidermal growth factor receptor 2 negative (HER2-)/Androgen receptor-positive (AR +) MBC with 1 to 3 previous treatments for metastatic disease
- Cohort 2: AR+/HR+/HER2 +/- Tumors: Postmenopausal women with hormone receptor (HR) positive (ER+ and/or PR+) /AR-positive (+) refractory MBC who have progressed after at least one and up to 3 previous hormonal treatments for metastatic disease.
Period: Overall Study
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Started | 27 (One participant was found to be ineligible after starting with study treatment and hence excluded from further analyses) | 44
Completed | 0 | 0
Not Completed | 27 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors | Total
Number analyzed (Participants) | 27 | 44 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (13.73) | 63.1 (11.34) | 61.1 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 44 | 71
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 23 | 43 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 22 | 39 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 44 | 71
Patients with Bone-only disease [Count of Participants; unit: Participants] | 4 | 8 | 12
HER2 positive patients [Count of Participants; unit: Participants] | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Response rate (RR) will be estimated as the percentage of patients exhibiting complete response or partial response out of all evaluable cases. Complete Response is defined per RECIST as the disappearance of all target/non-target lesions and normalization of tumor markers. Partial Response is defined per RECIST as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Complete and partial responses were confirmed at least 4 weeks after the initial response.
Time Frame: upto 36 months
Population: One participant in cohort 1 was found to be ineligible after starting treatment and was excluded from the analysis. Participants with bone-only metastases (4 in cohort 1 and 8 in cohort 2) were excluded from the analysis as they are not evaluable by RECIST V1.1. 14 participants, 1 in cohort 1 and 13 in cohort 2 who discontinued treatment prior to having a post-baseline scan were excluded. Participants who received at least one dose of study drug and with one post-baseline scan were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 21 | 23
percentage of participants | 4.8 [0.1 to 23.82] | 0 [0 to 14.82]

2. Primary Outcome: Disease Control Rate (DCR)
Description: Defined as the percentage of patients who do not exhibit progression (CR+PR+SD) at 6 months among those patients who are evaluable for response by RECIST V1.1. Complete Response is defined per RECIST as the disappearance of all target/non-target lesions and normalization of tumor markers. Partial Response is defined per RECIST as At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Stable disease is defined per RECIST as Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest (nadir) sum LD since the treatment started.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 21 | 23
percentage of participants | 4.8 [0.1 to 23.8] | 8.7 [1.1 to 28]

3. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events as a Measure of Safety
Description: Assessments will be made through analysis of the reported incidence of treatment-related Adverse Events as determined by the investigator and assessed by NCI CTCAE, Version 4.0.
Time Frame: weekly for 4 weeks then every 8 weeks until end of study treatment, up to 36 months.
Population: One participant in cohort 1 was found to be ineligible after starting treatment and hence was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
Participants | 20 | 38

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the first day of treatment until the day tumor progression or date of death was documented. The response was evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Every 8 weeks during treatment then every 6 months for 2 years, annually thereafter up to 5 years.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
months | 2 [1.2 to 5.2] | 1.8 [1.7 to 3.6]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the first treatment until the date of death due to any cause. In the absence of confirmation of death or lack of data beyond the follow-up period, the survival time was censored to the last date the participant was known to be alive.
Time Frame: After disease progression is documented, survival was monitored every 6 months for 2 years and annually thereafter up to 5 years.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
months | 10.2 [4.3 to NA] — The upper limit was not reached by the Kaplan-Meier method during the follow-up period due to an insufficient number of participants with events | 7.6 [3.9 to 9.7]

6. Secondary Outcome: Measurement of Serum Hormone Levels - Estradiol
Description: Blood samples collected At baseline, at day 1 of cycle 2 and 4, and at end of treatment visit to test for serum estradiol levels
Time Frame: At baseline, at day 1 of cycle 2 and 4 (treatment cycle repeated every 4 weeks), and at end of treatment visit, up to 36 months
Population: One participant in cohort 1 was found to be ineligible after starting treatment and hence was excluded from the analysis. Available data from the samples collected at each timepoint is reported.
Measure: Mean (Full Range); unit: pg/ml
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
pg/ml
  Baseline: number analyzed (Participants) | 26 | 41
  Baseline | 31.99 [5 to 235] | 29.16 [6 to 138]
  Cycle 2 Day 1: number analyzed (Participants) | 17 | 28
  Cycle 2 Day 1 | 22.29 [0 to 91] | 26.99 [7.6 to 143]
  Cycle 4 Day 1: number analyzed (Participants) | 7 | 6
  Cycle 4 Day 1 | 20.86 [0 to 70] | 33 [5 to 124]
  End of Treatment: number analyzed (Participants) | 17 | 33
  End of Treatment | 25.46 [5 to 144] | 28.15 [5 to 87]

7. Secondary Outcome: Measurement of Serum Hormone Levels - Total Testosterone
Description: Blood samples were collected at baseline, on day 1 of cycles 2 and 4, and at end of treatment visit to test total testosterone levels
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Full Range); unit: ng/dL
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
ng/dL
  Baseline: number analyzed (Participants) | 25 | 39
  Baseline | 16.36 [0 to 65] | 24.79 [2 to 404]
  Cycle 2 Day 1: number analyzed (Participants) | 17 | 27
  Cycle 2 Day 1 | 4.23 [0 to 11] | 4.35 [1 to 23]
  Cycle 4 Day 1: number analyzed (Participants) | 7 | 5
  Cycle 4 Day 1 | 3.71 [1 to 8] | 2.4 [1 to 4]
  End of Treatment: number analyzed (Participants) | 16 | 30
  End of Treatment | 6.11 [0 to 20] | 8.5 [0 to 42]

8. Secondary Outcome: Measurement of Serum Hormone Levels - Free Testosterone
Description: Blood samples were collected At baseline, at day 1 of cycle 2 and 4, and at end of treatment visit to test free testosterone levels
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
pg/mL
  Baseline: number analyzed (Participants) | 25 | 40
  Baseline | 1.62 [0.3 to 6.2] | 4.13 [0 to 111.3]
  Cycle 2 Day 1: number analyzed (Participants) | 14 | 23
  Cycle 2 Day 1 | 0.31 [0 to 0.7] | 0.39 [0.1 to 1.8]
  Cycle 4 Day 1: number analyzed (Participants) | 7 | 5
  Cycle 4 Day 1 | 0.36 [0.1 to 0.6] | 0.16 [0.1 to 0.3]
  End of treatment: number analyzed (Participants) | 15 | 28
  End of treatment | 0.6 [0 to 2] | 1.01 [0 to 3.7]

9. Secondary Outcome: Measurement of Serum Hormone Levels - Sex Hormone-binding Globulin
Description: Blood samples were collected at baseline, on day 1 of cycles 2 and 4, and at end of the treatment visit for sex hormone-binding globulin (SHBG) levels
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Full Range); unit: nmol/L
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
nmol/L
  Baseline: number analyzed (Participants) | 26 | 41
  Baseline | 81.95 [28 to 191.1] | 72.88 [23 to 162]
  Cycle 2 Day 1: number analyzed (Participants) | 18 | 28
  Cycle 2 Day 1 | 82.7 [25 to 183] | 91.93 [20 to 262]
  Cycle 4 Day 1: number analyzed (Participants) | 7 | 5
  Cycle 4 Day 1 | 67.17 [43 to 142.2] | 118.54 [68 to 168]
  End of Treatment: number analyzed (Participants) | 16 | 31
  End of Treatment | 77.69 [19 to 163] | 73.48 [21 to 190]

10. Secondary Outcome: Measurement of Serum Hormone Levels - Adrenocorticotropic Hormone
Description: Blood samples were collected at baseline, on day 1 of cycles 2 and 4, and at end of the treatment visit to test for adrenocorticotropic hormone (ACTH) levels
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Full Range); unit: pg/mL
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
pg/mL
  Baseline: number analyzed (Participants) | 24 | 36
  Baseline | 16.86 [4.9 to 41] | 18.61 [4 to 71]
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 23
  Cycle 2 Day 1 | 62.82 [4.3 to 189] | 58.04 [5 to 255]
  Cycle 4 Day 1: number analyzed (Participants) | 6 | 5
  Cycle 4 Day 1 | 56.55 [10.44 to 104.9] | 214.94 [8 to 845]
  End of treatment: number analyzed (Participants) | 18 | 27
  End of treatment | 42.14 [5 to 161] | 40.26 [5 to 265]

11. Secondary Outcome: Measurement of Serum Hormone Levels - Dehydroepiandrosterone Sulfate (DHEA-S)
Description: Blood samples were collected at baseline, on day 1 of cycles 2 and 4, and at end of the treatment visit dehydroepiandrosterone sulfate (DHEA-S) levels
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Full Range); unit: µg/dL
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
µg/dL
  Baseline: number analyzed (Participants) | 26 | 41
  Baseline | 74.63 [9 to 199] | 54.8 [9 to 146]
  Cycle 2 Day 1: number analyzed (Participants) | 18 | 27
  Cycle 2 Day 1 | 16.54 [2 to 43] | 14.48 [2 to 82]
  cycle 4 Day 1: number analyzed (Participants) | 7 | 5
  cycle 4 Day 1 | 23.29 [3 to 79] | 10.3 [2 to 25.5]
  End of Treatment: number analyzed (Participants) | 17 | 33
  End of Treatment | 36.85 [1 to 168] | 34.31 [2 to 158]

12. Secondary Outcome: Measurement of Serum Hormone Levels - Cortisol
Description: Blood samples to test for serum cortisol levels
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Full Range); unit: µg/dL
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 26 | 44
µg/dL
  Baseline: number analyzed (Participants) | 24 | 42
  Baseline | 10.45 [3.7 to 21.7] | 12.89 [4.2 to 31.1]
  Cycle 2 Day 1: number analyzed (Participants) | 18 | 28
  Cycle 2 Day 1 | 7.08 [2.3 to 13.7] | 6.91 [2 to 14.4]
  cycle 4 Day 1: number analyzed (Participants) | 7 | 4
  cycle 4 Day 1 | 7.14 [5.7 to 9.8] | 11 [3.9 to 24.9]
  End of Treatment: number analyzed (Participants) | 16 | 32
  End of Treatment | 8.16 [1.5 to 13.6] | 12.34 [1.7 to 42.7]

13. Other Pre Specified Outcome: Number of Participants With PTEN Gene Expression Status of Positive, Weak Positive, or Negative
Description: Archived tumor tissue was assayed for loss of phosphatase and tensin homolog (PTEN) biomarker. PTEN loss was determined by immunohistochemistry (IHC) staining. pTEN Positive by IHC is defined as strongly positive (2+ intensity) staining for PTEN protein expression in the entire tumor or the vast majority of the tumor cells. pTEN Negative by IHC is defined as no staining (0+intensity) in entire tumor cells for pTEN protein expression. pTEN Weakly positive(1+intensity) by IHC is defined as tumor cells showing weak pTEN protein expression.
Time Frame: At pre-screening
Population: Intent to treat analysis set. All enrolled participants' tissue was analyzed for loss of gene expression. Results are not reported for 6 participants in cohort 1, and 10 participants in cohort 2 who could not be assayed because of insufficient tissue available for testing or because their assay had indeterminate results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 20 | 34
Participants
  Positive | 6 | 18
  Weak Positive | 1 | 7
  Negative | 13 | 9

14. Other Pre Specified Outcome: Number of Participants With PIK3CA Gene Mutation Status of Mutated or No Mutation
Description: Archived tumor tissue was assayed for the phosphatidylinositol 3-kinase (PIK3CA) biomarker. PIK3CA hotspot mutations at codons 88, 539-549, 1020-1025, 1043-1049 were tested by pyrosequencing. 'PIK3CA-'mutated' is defined as the presence of mutation in one of the codons 88, 539-549, 1020-1025, 1043-1049 of the PIK3CA gene.
  PIK3CA-'no mutation' is defined as the absence of mutation in codons 88, 539-549, 1020-1025, 1043-1049 of the PIK3CA gene.
Time Frame: At pre-screening
Population: Intent to treat analysis set. All enrolled participants' tissue was analyzed for loss of gene expression. Results are not reported for 8 participants in cohort 1, and 11 participants in cohort 2 who could not be assayed because of insufficient tissue or because of their assay had indeterminate results.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
Number analyzed (Participants) | 18 | 33
Participants
  Mutated | 3 | 12
  No mutation | 15 | 21

ADVERSE EVENTS:
Time Frame: Up to 36 months for Serious Adverse Events and Other Adverse Events. Up to 5 years for All-Cause Mortality.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from the day of the first dose to 30 days after the last dose of the study medication and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
  One participant in cohort 1 was found to be ineligible after starting with study treatment and hence excluded from further analyses.
Groups:
- Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors: Patients with estrogen receptor-negative (ER-)/progesterone receptor negative (PR-)/ human epidermal growth factor receptor 2 negative (HER2-)/AR-positive (+) MBC with 1 to 3 previous treatments for metastatic disease
Arm/Group | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors | Cohort 2: AR+/HR+/HER2 +/- Tumors
All-Cause Mortality (participants affected / at risk) | 23/26 | 39/44
Serious Adverse Events (participants affected / at risk) | 11/26 | 11/44
Other Adverse Events (participants affected / at risk) | 20/26 | 38/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors (N=26) | Cohort 2: AR+/HR+/HER2 +/- Tumors (N=44)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial mass (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Patients With AR+/ER-/PR-/HER2- Tumors (N=26) | Cohort 2: AR+/HR+/HER2 +/- Tumors (N=44)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 3 (3)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (5)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 3 (4)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Eyelid margin crusting (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 5 (7)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (8) | 12 (14)
Dental paraesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip exfoliation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (15) | 19 (24)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 10 (14)
Asthenia (General disorders) | 0 (0) | 3 (3)
Chest pain (General disorders) | 0 (0) | 2 (2)
Chills (General disorders) | 2 (2) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 13 (16) | 21 (34)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 1 (3)
Malaise (General disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 3 (3) | 3 (4)
Pain (General disorders) | 3 (3) | 3 (3)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1)
Tenderness (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 5 (5)
Amylase (Investigations) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 3 (5) | 3 (7)
Aspartate aminotransferase (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (6) | 6 (7)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (6) | 4 (5)
Blood bilirubin increased (Investigations) | 0 (0) | 5 (7)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 1 (3) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 2 (3) | 0 (0)
Haemoglobin (Investigations) | 0 (0) | 1 (3)
Haemoglobin decreased (Investigations) | 1 (3) | 0 (0)
Lipase (Investigations) | 0 (0) | 2 (3)
Lipase increased (Investigations) | 2 (6) | 6 (11)
Neutrophil count (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count (Investigations) | 0 (0) | 1 (4)
Platelet count decreased (Investigations) | 2 (4) | 3 (4)
Protein total increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 5 (5)
White blood cell count (Investigations) | 0 (0) | 1 (2)
White blood cell count decreased (Investigations) | 2 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (8)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (7) | 10 (13)
Horner's syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 2 (5) | 3 (3)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (4)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 6 (6) | 4 (4)
Hypertension (Vascular disorders) | 3 (8) | 6 (10)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT01990209/Prot_SAP_000.pdf